CLINICAL TRIAL: NCT00978952
Title: Large Diameter Advanta™ V12 Covered Stent Trial for Coarctation of the Aorta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atrium Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 803
Record Dates: First submitted 2009-09-14; First posted 2009-09-17 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Coarctation of the Aorta
MeSH Terms: conditions — Aortic Coarctation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Investigational Group (Experimental): Use of Large Diameter Advanta™ V12 Covered Stent.
  Interventions: Device: Large Diameter Advanta™ V12 Covered Stent

INTERVENTIONS:
Device: Large Diameter Advanta™ V12 Covered Stent — Stent placement

SUMMARY:
This study is designed as a prospective, multicenter, non-randomized, single arm study to assess the safety and effectiveness of the Large Diameter Advanta™ V12 Covered Stent for stent implantation in coarctations of the aorta.

DETAILED DESCRIPTION:
The performance metric for comparison is based on data from the Congenital Cardiovascular Interventional Study Consortium (CCISC) as reported by Golden and Hellenbrand [1]. The CCISC experience from 1989 to 2005 shows a true procedural success rate of 98.6%.

The patient population will be subjects with coarctation of the aorta. A total of 70 subjects, children, adolescents and adults, will be enrolled at up to 15 study sites. Baseline clinical and angiographic assessment will determine the subject's eligibility for enrollment in the study. Subjects will continue in the study for long term annual follow-up through 3, 4, and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a presence of native or recurrent coarctation of the aorta as confirmed by blood pressure gradient, 2D-echocardiography with Doppler or angiography.
* Subject weighs a minimum of 30 kg.
* The peak pressure gradient is ≥20 mmHg systolic blood pressure across the coarctation site.
* Vessels at access site can accept a minimum size of 9 French for a 12 mm balloon and 11 French for a 14 and 16 mm balloon.
* Coarctation can be successfully crossed with a guide wire, sheath and device.
* Diameter of transverse arch distal to left subclavian artery is between 9.5 mm and 20 mm in diameter.
* Subject is able and willing to adhere to all required follow-up visits and testing.
* Subject is able and willing to adhere to the required follow-up medication regimen.

Exclusion Criteria:

* The physician is not able to access the coarctation with standard techniques.
* Presence of other thoracic aortic arterial lesions or aneurysms requiring treatment within 30 days of the implant procedure.
* Length of coarctation is greater than 45 mm in length.
* Connective tissue and genetic disorders, including William, Marfan, Turner, Noonan syndrome.
* The coarctation has adjacent, acute thrombus.
* The coarctation was previously treated with a stent.
* Proximity of the coarctation to an important side branch resulting in crossing of the side branch with the Large Diameter Advanta™ V12 Covered Stent device (e.g. "jailing" of the branch vessel).
* Subject has a tubular graft, interposition graft, stent graft at or near the coarctation site that would be interfere with delivery, positioning, expansion or stabilization of the Large Diameter Advanta™ V12 Covered Stent
* Subject has contrast agent hypersensitivity that cannot be adequately premedicated, has a hypersensitivity to stainless steel, expanded polytetrafluoroethylene (ePTFE) or has intolerance to antiplatelet, anticoagulant, or thrombolytic medications.
* Bloodstream infection
* Subject is pregnant or breastfeeding.
* Subject has a co-morbid illness that may result in a life expectancy of less than 1 year.
* The investigator deems the subject to be an inappropriate candidate for the study.
* Subject is participating in an investigational study of a new drug, biologic or device at the time of study screening. NOTE: Subjects who are participating in the long term follow-up phase of a previously investigational and now approved product are not excluded by this criterion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-09; Primary Completion 2013-05 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy | 12 month
  The mean difference between Diastolic Velocity (DV)/Systolic Velocity(SV) pre and post procedure (i.e. pre procedure DV/SV - post procedure DV/SV) minus the difference between 12 month and post procedure (i.e. 12 month DV/SV - post procedure DV/SV).
Primary Safety | 30 days of procedure
  30 day morbidity rate of Major Adverse Events (MAE)and Major Adverse Vascular Events (MAVE)

SECONDARY OUTCOMES:
Secondary Safety | procedural (time zero)
  Device success, defined as the successful delivery and deployment of the study stent and intact retrieval of the delivery system.
Secondary Safety | 12 month
  No post procedural stent migration, where migration is defined as displacement of the stent >20mm from an established anatomical landmark verified during deployment.
Secondary Safety | 12 months
  Major Adverse Events (MAE)and Major Adverse Vascular Events (MAVE)

CONTACTS AND LOCATIONS:
Overall Officials: Elchanan Bruckheimer, MD, Principal Investigator — Schneider Children's Medical Center, Israel
Locations (9):
- The Children's Hospital at Westmead, Sydney, Australia
- Instituto Dante Pazzanese de Cardiologia, São Paulo, Brazil
- Hospital for Sick Children Labatt Family Heart Centre, Toronto, Ontario, Canada
- Germany (3):
  - Heart Institute Berlin, Berlin
  - CardioVascular Center, Frankfurt
  - Asklepios Klinik Sankt Augustin, Sankt Augustin
- Schneider Children's Medical Center, Petah Tikva, Israel
- San Donato Hospital, Milan, Italy
- Bristol Royal Hospital for Children and Bristol Royal Infirmary, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bruckheimer E, Birk E, Benson L, Butera G, Martin R, Roberts PA, Schneider MBE, Schubert S, Sievert H, Pedra CCA. Large Diameter Advanta V12 Covered Stent Trial for Coarctation of the Aorta: COARC Study. Circ Cardiovasc Interv. 2021 Dec;14(12):e010576. doi: 10.1161/CIRCINTERVENTIONS.121.010576. Epub 2021 Nov 9. PMID 34749516